CLINICAL TRIAL: NCT04429607
Title: Treatment of Sebaceous Hyperplasia With PDL and Nd:YAG Versus Erbium:YAG: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor of Dermatology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00211739
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Sebaceous Hyperplasia
MeSH Terms: interventions — Lasers, Dye; Curettage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Erbium:YAG Laser (Active Comparator): Solitary lesions will be randomized to a group, thus, a patient may receive all three treatments, each on different lesions. Patients will undergo two total treatment sessions at 2-6 week intervals.
  Interventions: Device: Erbium:YAG Laser
- PDL plus Nd:YAG (Active Comparator): Solitary lesions will be randomized to a group, thus, a patient may receive all three treatments, each on different lesions. Patients will undergo two total treatment sessions at 2-6 week intervals.
  Interventions: Device: Pulsed Dye Laser; Device: Nd:YAG Laser
- ED&C treatment (Active Comparator): Solitary lesions will be randomized to a group, thus, a patient may receive all three treatments, each on different lesions. Patients will undergo two total treatment sessions at 2-6 week intervals.
  Interventions: Procedure: Electrodessication and curettage

INTERVENTIONS:
Device: Erbium:YAG Laser — Erbium:YAG 2940nm will be performed using single spot, multiple pulses on lesions.
  Arms: Erbium:YAG Laser
Device: Pulsed Dye Laser — PDL will be performed using settings of 6-10 J/s2 on lesions.
  Other Names: PDL
  Arms: PDL plus Nd:YAG
Device: Nd:YAG Laser — Nd:YAG 1064nm will be performed using settings of 60-110 J/s2 on lesions.
  Arms: PDL plus Nd:YAG
Procedure: Electrodessication and curettage — Electrodessication and curettage will be performed using an epilating needle, followed by curettage on lesions.
  Other Names: ED&C
  Arms: ED&C treatment

SUMMARY:
The purpose of this study is to compare treatment of sebaceous hyperplasia with pulsed dye laser (PDL) plus neodymium doped yttrium aluminum garnet laser (Nd:YAG) versus erbium doped yttrium aluminum garnet (erbium:YAG) laser versus electrodesiccation and curettage (ED&C).

This is a randomized clinical trial. Approximately 18 participants will enrolled. Each participant will have their sebaceous hyperplasia lesions randomized to receive either Erbium:YAG, PDL plus Nd:YAG, or ED&C treatment. Solitary lesions will be randomized to a group, thus, a patient may receive all three treatments, each on different lesions. Lesions will be treated twice, 2-6 weeks after the first treatment. Lesion size and count will be measured before treatment and at follow-up 4-12 weeks after the first treatment. This study is a pilot study designed to determine the feasibility of these procedures.

Subjects currently living in the Chicago metropolitan area and meet inclusion/exclusion criteria will be considered for enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. Receiving cosmetic treatment for sebaceous hyperplasia
3. In good general health as assessed by the investigator
4. Participants must have the ability to understand and the willingness to sign a written informed consent prior to registration on study

Exclusion Criteria:

1. Patient pregnant or nursing
2. Patient with history of poor wound healing that would result in hypertrophic scar or keloid at the discretion of the physician
3. Patient with recent sun exposure that would result in pigment changes at the discretion of the physician
4. Subject unwilling to sign an IRB approved consent form
5. Participants who are unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in size of sebaceous hyperplasia | 4-12 weeks
  Change in size of sebaceous hyperplasia from baseline to 4-12 weeks after first treatment by measuring length and width in mm of each lesion.
Change in sebaceous hyperplasia lesion count | 4-12 weeks
  Change in sebaceous hyperplasia lesion count from baseline to 4-12 weeks after first treatment

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No